CLINICAL TRIAL: NCT02433431
Title: Mechanisms of Mindfulness and Stress Resilience: A Mobile App Mindfulness Training Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Collaborators: Mind and Life Institute, Hadley, Massachusetts (Other); Yoga Science Foundation (Other); Penn State University (Other); University of Pittsburgh (Other); Virginia Commonwealth University (Other); 01 Expert Systems, LLC (Industry)
Responsible Party: Principal Investigator, Emily Lindsay, Doctoral Student, Carnegie Mellon University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRBSTUDY2015_00000122
Record Dates: First submitted 2015-04-23; First posted 2015-05-05 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Psychological Stress; Mindfulness
Keywords: mindfulness; psychological stress; immune marker; wellness programs; mobile applications; cortisol
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mindfulness Training (Active Comparator): 14-lesson audio-guided mindfulness training program instructing present-moment attention and an orientation of acceptance
  Interventions: Behavioral: Mindfulness Training
- Mindful Attention Only Training (Active Comparator): 14-lesson audio-guided mindfulness training program instructing present-moment attention only
  Interventions: Behavioral: Mindful Attention Only Training
- Analytic Thinking Training (Active Comparator): 14-lesson audio-guided analytic thinking program encouraging reflection on one's thoughts, feelings, and behaviors, but not instructing mindfulness
  Interventions: Behavioral: Analytic Thinking Training

INTERVENTIONS:
Behavioral: Mindfulness Training — Mindfulness training intervention consisting of 14 x 20-minute audio-guided lessons that participants access on their smartphones during the 14-day intervention period.
  Arms: Mindfulness Training
Behavioral: Mindful Attention Only Training — Mindful attention training intervention consisting of 14 x 20-minute audio-guided lessons that participants access on their smartphones during the 14-day intervention period.
  Arms: Mindful Attention Only Training
Behavioral: Analytic Thinking Training — Comparison analytic thinking intervention consisting of 14 x 20-minute audio-guided lessons that participants access on their smartphones during the 14-day intervention period.
  Arms: Analytic Thinking Training

SUMMARY:
The purpose of this study is to test the active components of mindfulness meditation for reducing psychological stress and improving biomarkers of health. This study compares the effects of three brief trainings: (1) training in both present-moment attention and mindful acceptance, (2) training in present-focused attention, and (3) an active psychological training with no mindfulness content.

DETAILED DESCRIPTION:
Mindfulness meditation practices are widely used among the general public, with people seeking to reduce stress, pain, inflammation, depression, and disease symptoms. Moreover, randomized controlled trials have shown mindfulness training programs to be effective in improving a broad range of psychological and physical health outcomes, particularly among populations with high stress burdens. Still, little is known about the mechanisms underlying mindfulness training that drive these effects. This study tests the active components of mindfulness that impact stress responding and health biomarkers.

The study separates attention and acceptance mindfulness instructions into three 14-day training programs delivered to a stressed adult population: (1) attention and acceptance instructions, (2) attentional monitoring instructions only, or (3) analytic thinking with no mindfulness instruction. Intervention programs are delivered on participants' own smartphones, providing a platform for maximal experimental control in testing the active ingredients of mindfulness training.

Participants are recruited from the Pittsburgh community. At a baseline laboratory session, they complete psychosocial questionnaires and tasks and provide a dried blood spot sample. On their own, they complete pre- and post-intervention Ecological Momentary Assessment measures of stress, attention, and acceptance in daily life. Between these assessments, participants have 14 days to complete their randomly assigned 14-lesson intervention program. Participants return to the lab for post-intervention assessments (questionnaires, tasks, dried blood sample), listen to a final training session from their intervention program, and complete the Trier Social Stress Test. Participants are compensated.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Moderate- to high-stress (4-item Perceived Stress Scale score of 6 or higher)

Exclusion Criteria:

* Diagnosis of chronic mental (e.g., recurrent depression, schizophrenia, personality disorder) or physical disease (e.g., cancer, HIV, heart disease, diabetes, bleeding disorder)
* Hospitalization in past 3 months
* Medication use that interferes with HPA-axis activity (e.g., corticosteroids)
* Current oral contraceptive use
* Current antibiotic, antiviral, or antimicrobial treatment
* Travel outside the country within the past 6 months to any country on the CDC travel alert list
* Recreational drug use, excessive alcohol or tobacco use
* Significant experience with or daily practice of mindfulness meditation or related mind-body practice

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2015-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Daily life stress assessed via Ecological Momentary Assessment | change from baseline 3-day period to post-intervention 3-day period, which is an average of 2.5 weeks
Inflammatory Biomarkers assessed via Dried Blood Spot | change from baseline to post-intervention, which is an average of 3.5 weeks
  Five Dried Blood Spot samples are obtained from participants' finger for assessment of circulating markers of inflammation (CRP, IL-6).

SECONDARY OUTCOMES:
Daily life state attention and acceptance assessed via Ecological Momentary Assessment | change from baseline 3-day period to post-intervention 3-day period, which is an average of 2.5 weeks
Subjective stress in response to social evaluative threat (TSST) | assessed at post-intervention, which is an average of 3.5 weeks
Salivary Cortisol AUC in response to social evaluative threat (TSST) | assessed at post-intervention, which is an average of 3.5 weeks, at time 0, and 25, 35, and 60 minutes post-TSST
Blood Pressure reactivity to social evaluative threat (TSST) | assessed at post-intervention, which is an average of 3.5 weeks, at 2-minute intervals during session
Evening salivary cortisol | change from baseline 3-day period to post-intervention 3-day period, which is an average of 2.5 weeks
Sustained attention measured by the Dichotic Listening Task | change from baseline to post-intervention, which is an average of 3.5 weeks

OTHER OUTCOMES:
Daily life affect assessed via Ecological Momentary Assessment | change from baseline 3-day period to post-intervention 3-day period, which is an average of 2.5 weeks
Daily life social interactions assessed via Ecological Momentary Assessment | change from baseline 3-day period to post-intervention 3-day period, which is an average of 2.5 weeks
Perceived stress measured by the PSS | change from baseline to post-intervention, which is an average of 3.5 weeks
Mindfulness facets measured by the FFMQ-sf | change from baseline to post-intervention, which is an average of 3.5 weeks
Mindfulness measured by the PHLMS | change from baseline to post-intervention, which is an average of 3.5 weeks
Attentional control measured by the ACS | change from baseline to post-intervention, which is an average of 3.5 weeks
Nonattachment measured by Nonattachment Scale | change from baseline to post-intervention, which is an average of 3.5 weeks
Subjective health measured by the SF-12 | change from baseline to post-intervention, which is an average of 3.5 weeks
Sleep quality measured by the PSQI-sf | change from baseline to post-intervention, which is an average of 3.5 weeks
Loneliness measured by the UCLA Loneliness Scale | change from baseline to post-intervention, which is an average of 3.5 weeks
Interpersonal support measured by the ISEL-12 | change from baseline to post-intervention, which is an average of 3.5 weeks
Social network measured by the SNI | change from baseline to post-intervention, which is an average of 3.5 weeks
Depression measured by the CES-D-10 | change from baseline to post-intervention, which is an average of 3.5 weeks
Mind-wandering measured by the RRQ | change from baseline to post-intervention, which is an average of 3.5 weeks
Treatment expectancies measured by Credibility/Expectancy Questionnaire | post-intervention, which is an average of 3.5 weeks
Alerting, orienting, and executive control measured by the ANT task | post-intervention, which is an average of 3.5 weeks
Subjective responses to the training program intervention | composite of ratings made after each of 14 intervention lessons, an average of 2 weeks following baseline

CONTACTS AND LOCATIONS:
Overall Officials: Emily K Lindsay, MS, Principal Investigator — Carnegie Mellon University; J. David Creswell, PhD, Principal Investigator — Carnegie Mellon University
Locations (1):
- Carnegie Mellon University, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Lindsay EK, Young S, Creswell JD. Mindfulness training fosters a positive outlook during acute stress: A randomized controlled trial. Emotion. 2025 Jun;25(4):815-826. doi: 10.1037/emo0001452. Epub 2024 Nov 21. PMID 39570681
- [Derived] Lindsay EK, Chin B, Greco CM, Young S, Brown KW, Wright AGC, Smyth JM, Burkett D, Creswell JD. How mindfulness training promotes positive emotions: Dismantling acceptance skills training in two randomized controlled trials. J Pers Soc Psychol. 2018 Dec;115(6):944-973. doi: 10.1037/pspa0000134. PMID 30550321